CLINICAL TRIAL: NCT05530434
Title: Transpulmonary Pressure Guided Weaning From Invasive Mechanical Ventilation in Obese Patients With Respiratory Failure
Brief Title: Transpulmonary Pressure Guided Mechanical Ventilation Weaning in Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Meredith E. Sloan, Instructor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMMC-IRB-2022-301
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Failure; Obesity
Keywords: Transpulmonary pressure; Respiratory failure; Obesity; Invasive mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transpulmonary pressure guided positive end expiratory pressure (Experimental): Patients in this group will have the positive end expiratory pressure on the ventilator set to a transpulmonary pressure of 0-2 cm H2O during ventilation and spontaneous breathing trials.
  Interventions: Other: transpulmonary pressure guided positive end expiratory pressure
- Standard positive end expiratory pressure (Active Comparator): Patients in this groups will have the positive end expiratory pressure on the ventilator set by the clinician during ventilation and set to a standard positive end expiratory pressure of 5-8 cm H2O during spontaneous breathing trials.
  Interventions: Other: standard positive end expiratory pressure

INTERVENTIONS:
Other: transpulmonary pressure guided positive end expiratory pressure — Positive end expiratory pressure will be titrated to achieve a transpulmonary pressure of 0-2 cm H2O
  Arms: Transpulmonary pressure guided positive end expiratory pressure
Other: standard positive end expiratory pressure — Positive end expiratory pressure will be set to a standard 5-8 cm H2O by the clinician for spontaneous breathing trials
  Arms: Standard positive end expiratory pressure

SUMMARY:
This study will look at whether accounting for the amount of pressure generated by the chest wall and abdomen in a obese patient, using a measurement called transpulmonary pressure, can help shorten the amount of time patients spend on the ventilator. By decreasing the amount of time patients spend on the ventilator, they are less likely to develop complications such as infections, weakness or more procedures.

DETAILED DESCRIPTION:
Managing obese patients on the ventilator can be difficult due to the changes in their respiratory mechanics with little evidence as to best practices. This research will assess the utility of transpulmonary pressures in guiding mechanical ventilation in obese patients. This study with specifically look at whether using transpulmonary pressure guided positive end expiratory pressure (PEEP) titration for ventilation and spontaneous breathing trials (SBT) will shorten the time to liberation for obese patients on invasive mechanical ventilation for respiratory failure. The transpulmonary pressures will be calculated daily for all patients. Patients will also be assessed daily for readiness for SBT. In the intervention group, subjects' PEEP will be titrated to achieve an end expiratory transpulmonary pressure of 0-2 cm H2O. This PEEP will be used for the SBT and clinicians will be encouraged to keep their patients on this PEEP after the SBT if they are not extubated. In the control group, patients will also be assessed daily for SBT readiness but will be managed with standard set pressures of 5 to 10 cm H2O of PEEP and 5 to 8 cm H2O of pressure above PEEP. The primary team can perform a T piece trial prior to extubation as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* on invasive mechanical ventilation for respiratory failure for < 48 hours
* obese class II or higher (BMI greater than or equal to 35.0 kg/m2)

Exclusion Criteria:

* contraindications to esophageal balloon catheter placement including esophageal, nasofacial, gastrointestinal abnormalities and platelets <10,000/microliter
* known pleural disease such as persistent pneumothorax, pleural effusion, or pleurodesis
* neuromuscular disease
* requires chronic mechanical ventilation prior to enrollment
* severe neurologic injury
* known difficult airway
* life expectance is less than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Ventilator free days | 30 days
  Number of ventilator free days

SECONDARY OUTCOMES:
Mortality | 30 days
  Number of patients who died during the study
Days on invasive mechanical ventilation | 30 days
  Number of days patient spent on mechanical ventilation
Re-intubation rate | 30 days
  Percentage of patients who were re-intubated after extubation failure
Number of tracheostomies | 30 days
  Number of patients who received tracheostomies
PEEP at extubation | 30 days
  the amount of positive end expiratory pressure set on the ventilator prior to extubation
Intensive care unit length of stay | 30 days
  Number of days spent in the intensive care unit
Hospital length of stay | 30 days
  Number of days spent in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No